CLINICAL TRIAL: NCT00003837
Title: Compound 506U78 (NSC 686673) in Patients With Relapsed or Refractory T-Cell ALL or T-Cell Lymphoblastic Lymphoma
Brief Title: 506U78 in Treating Patients With Relapsed or Refractory T-cell Acute Lymphoblastic Leukemia or T-cell Lymphoblastic Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066994; CTEP-TRC-9701; CWRU-TRC-1499
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2005-12

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent adult acute lymphoblastic leukemia; T-cell adult acute lymphoblastic leukemia; recurrent adult lymphoblastic lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — nelarabine

INTERVENTIONS:
Drug: nelarabine

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Clinical trial to study the effectiveness of 506U78 in treating patients who have relapsed or refractory T-cell acute lymphoblastic leukemia or T-cell lymphoblastic lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Provide an investigational agent, 506U78, to physicians for the management of individual patients with relapsed or refractory T-cell acute lymphoblastic (lymphocytic) leukemia or T-cell lymphoblastic lymphoma who are not candidates for entry onto ongoing research clinical trials of higher priority.
* Evaluate the toxic effects of 506U78 when administered as a 2 hour IV infusion 3 days a week every 21 days in these patients.
* Evaluate the antitumor efficacy of this regimen in terms of rate of complete responses in these patients.

OUTLINE: Patients receive 506U78 over 2 hours on days 1, 3, and 5. Treatment repeats every 21 days for a maximum of 12 courses in the absence of unacceptable toxicity or disease progression.

Patients are followed every 3 months for one year and then every 6 months until death.

PROJECTED ACCRUAL: A minimum of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed relapsed or refractory T-cell acute lymphoblastic leukemia or T-cell lymphoblastic lymphoma

  * Tumor cells should exhibit phenotypic characteristics of these diseases
* No CNS involvement requiring intrathecal or craniospinal radiotherapy
* Must not be eligible for Intergroup, Cooperative Group, or local research studies of higher priority

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-3 OR
* Karnofsky 40-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 2.0 mg/dL

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 50 mL/min

Other:

* No neuropathy grade 2 or higher
* No history of significant neurological toxicity (grade 2 or greater) associated with prior chemotherapy or radiotherapy
* No active seizure disorder
* No active infection
* No other active concurrent malignancy except curatively treated basal cell carcinoma or carcinoma in situ of the cervix
* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior bone marrow transplantation allowed
* No concurrent allogeneic bone marrow transplantation

Chemotherapy:

* At least 3 weeks since prior chemotherapy (6 weeks for nitrosourea or mitomycin) and recovered
* No prior 506U78

Endocrine therapy:

* No concurrent systemic steroid therapy

Radiotherapy:

* See Disease Characteristics
* Prior radiotherapy allowed

Surgery:

* Not specified

Other:

* No other concurrent investigational therapy
* No concurrent treatment for seizures

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1999-09; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Provide an investigational agent to physicians for patients who are not candidates for entry onto ongoing research clinical trials of higher priority

SECONDARY OUTCOMES:
Toxicity
Antitumor efficacy as defined by the rate of complete hematologic responses

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J. Murgo, MD, Study Chair — NCI - Investigational Drug Branch
Locations (7):
- United States (7):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - NCI - Pharmaceutical Management Branch, Bethesda, Maryland
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania